CLINICAL TRIAL: NCT02339012
Title: The Genetic and Epigenetic Signatures of Translational Aging Laboratory Testing (GESTALT)
Brief Title: Genetic and Epigenetic Signatures of Translational Aging Laboratory Testing (GESTALT)
Status: Recruiting | Type: Observational
Sponsor: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 150063; 15-AG-0063
Record Dates: First submitted 2015-01-14; First posted 2015-01-15 (Estimated); Last update posted 2026-01-16 (Actual); Status verified 2025-12-10

CONDITIONS: Healthy Volunteers; Non-Healthy/Non-Frail; Frail
Keywords: Genome Wide Association; Biomarkers; Methylation; Phenotype; Cytometry; Natural History

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Frail: frail individuals ages 50-64 years; 65-79 years; 80+ years
- Healthy: healthy individuals ages 20-34 years; 35-39 years; 50-64 years; 65-79 years; 80+ years
- Non-Healthy/Non-Frail: non-healthy/non-frail individuals ages 20-34 years; 35-39 years; 50-64 years; 65-79 years; 80+ years

SUMMARY:
Background:

- Biomarkers are substances in people s blood and tissues. They help researchers understand diseases and signs of aging. Scientists want to do more research on biomarkers to find ways to improve quality of life in old age.

Objective:

- To learn more about biomarkers and their relationship to aging.

Eligibility:

- Adults at least 20 years old who weigh at least 110 pounds and have a body mass index below 30. They must agree that their genetic samples can be collected, studied, and stored.

Design:

* Participants will be screened with medical history, physical exam, EKG and blood and urine tests.
* Participants will have 3-day visits. They will return every 2 years.
* All visits include:
* Blood and urine collection
* Physical performance tests
* Health questionnaires
* Memory and problem-solving tests
* Magnetic Resonance Imaging (MRI) and Computerized Tomography (CT) scans.
* Muscle metabolism/ exercise tests
* Taste strips
* Muscle and/or skin biopsies/ red light therapy
* Retinal imaging/ eye tracking
* Sleep study
* ODD visits also include:
* Cytapheresis
* Bone marrow aspirate
* EVEN visits also include:
* Hyperglycemic CLAMP
* Lumbar Puncture (LP)
* Continuous Glucose Monitor (CGM)

DETAILED DESCRIPTION:
Under the assumption that aging is caused by dysfunction of specific biological mechanisms, it is reasonable to hypothesize that slowing aging should delay the onset of chronic diseases that typically affect older persons and improve their longevity and quality of life. Indeed, there is emerging evidence that factors associated with premature mortality are also involved in multiple pathologic conditions typical of aging. There is evidence that the study of aging and longevity requires a more comprehensive analysis of biological, environmental and phenotypic changes that occur with aging and how they are reflected by circulating and tissue biomarkers. A major limitation in this approach to date is that most studies of biomarkers rely on blood specimens, which may not recapitulate the biology of other tissues. In addition, although all cell types from the same person have exactly the same genetic code; information on epigenetic modifications, RNAm, and protein expression likely differ across cell types and at different points in time. Thus, global measures of these biomarkers in specific cell types can be affected by percentages of these cell types in the blood, and it is well known that such percentages change with aging and chronic diseases. More recently single cell biomarker assessment overcome such limitation and will be introduced in GESTALT in parallel with the measures already obtained.

In GESTALT, we will use cytapheresis to collect large number of PBMCs in the H group and we will draw blood to collect PBMCs in the NHF and F individuals dispersed over a wide age- range. The collection of large number of PBMCs is essential to obtain enough cells for each cell type to support measurements of the biomarkers of interest.

The information collected will be used to identify biomarkers that change with aging in healthy, non-healthy-or-frail and frail individuals, independent of changes in specific PBMCs cell types. We will also develop a statistical model that can be used by other studies of biomarkers to adjust their analysis for PBMCs cell type composition without having to perform complex and expensive measures, such as flow cytometry. The data collected in PBMCs will be compared to similar biomarker data obtained from muscle/fat and skin biopsies to understand to what extent biomarkers measured in the blood recapitulate similar changes that occur in different human tissues. Finally, once methodological limitations of measuring biomarkers in the blood have been addressed, we plan to assess the relationship of biomarkers assessed in specific circulating cell types, in the whole blood, bone marrow aspirate and in muscle/fat and skin biopsies to physiological measures that typically change with aging, including measures of body composition (anthropometrics, CT scan and MRI), energetics (spirometry at rest and during different degrees of exercise intensity), homeostatic equilibrium (hormones and inflammatory markers), neurological function (neurocognitive testing, brain MRI, nerve conduction studies). At even visits, we will focus on in depth characterization of phenotypes that are relevant for aging. Additionally, a modified schedule of testing will occur starting at Year 8. Year 8 Visit 4.5, which is between visits 4 and 5 and Year 18 Visit 8.5, which is between visits 8 and 9 and every 10 years thereafter. This strategy reduces the burden to participants but still allows delineating trajectories of essential variables and relate them longitudinally. The final goal is to develop new hypotheses about the biological nature of the aging process and how aging is associated with decline of physical and cognitive function.

ELIGIBILITY:
* Since the study of gene expression and epigenetic regulation are essential aims of GESTALT, all participants are required to consent to DNA/RNA testing and storage at all visits. Participants that refuse genetic testing and storage will not be eligible to participate or to continue to participate in the study.

The criteria below for each group pertains only to the Screening and Baseline Visits, except where otherwise noted. If any of the conditions develop while the participant is in the study, the participant remains in the study. However, participants that develop severe cognitive problems and are diagnosed by the cognition group with dementia, will no longer be able to participate in the study.

INCLUSION CRITERIA for the Healthy Group:

* Age greater than or equal to 20 years of age.
* Are willing to return every 2 years for study visit procedures.
* Agree to genetic (DNA/RNA) sample collection, analysis and storage.
* Have good venous access for cytapheresis and are in good health as determined by the Apheresis Health History Questionnaire and are found eligible for apheresis (Apheresis Eligibility form).
* Weigh greater than or equal to 110lbs and a body mass index (BMI) < 30.
* Do not have established genetic diseases such as sickle cell, hemochromatosis (iron overload), cystic fibrosis or Ehlers-Danlos syndrome (connective tissue disorder).
* Do not have autoimmune diseases such as Hashimoto's thyroiditis, Myasthenia Gravis or Rheumatoid arthritis.
* Report that they are able to perform daily self- care without assistance.
* Report that they able to walk independently for at least 400 meters without assistance and without developing severe symptoms.
* Report they are able to perform normal activities of daily living without shortness of breath (walking or climbing stairs) or other severe symptoms.
* Do not have cognitive impairment based on mental status screening tests and evaluations and in the absence of any drug treatment.
* Do not have a history of cardiovascular disease or cerebrovascular disease including angina (requiring treatment), myocardial infarction, congestive heart failure, uncontrolled hypertension, pacemaker, stroke, or transient ischemic attacks (TIA).
* Do not have a history of diabetes (requiring any medical treatment other than diet and exercise) and their fasting Glucose is <126 mg/dL.
* Do not have active (any activity in the last 10 years) cancer, except for locally limited squamous and basal cell cancer.
* Do not have clinically significant hormonal dysfunction (Self-reported or laboratory values out of range. Mild hypothyroidism in participants over 60 is not considered exclusion).
* Do not have a history of neurological diseases or birth defects (other than minor anatomical abnormalities, which do not affect physical and/or cognitive function).
* Do not have a history of kidney or liver disease (associated with reduced kidney or liver function).
* Do not have a history of severe gastrointestinal (G.I.) diseases, with symptoms or requiring chronic treatment such as gastroesophageal reflux disease (GERD), Crohn s disease or ulcerative colitis.
* Do not have a history of severe pulmonary disease such as chronic obstructive pulmonary disease (COPD) or asthma requiring continuous medication use.
* Do not have muscle-skeletal conditions due to diseases or traumas (that cause pathological weakness and/or chronic pain).
* Do not have a history of severe psychiatric conditions associated with behavioral problems or requiring absolute and continuous need for medical treatment.
* Do not have any medical condition that requires absolute and continuous need for long term treatment with antibiotics, corticosteroids, immunosuppressors, H2 blockers and/or proton pump inhibitors, or pain medications.
* Do not have a medical condition that requires the use of chronic anticoagulant medication such as Coumadin, heparin, or antiplatelet agents other than low dose aspirin.
* Do not have important sensory deficits (legally blind and/or any condition that precludes the participant from being tested with standard neuropsychological tests or providing informed consent).
* Are able to read and speak English.
* Are able to understand the study risks and procedures, and consent to participate in the study.
* Not currently pregnant or a nursing mother.
* Do not currently smoke and have not smoked in the past 3 months.
* Veins are adequate for cytapheresis.
* No current illness that as judged by the study physician substantially increases the risks associated with cytapheresis (active infections, allergies, etc.).
* No history of allergy to acid- citrate- dextrose (ACD) anticoagulant.
* No history of an active bleeding disorder such as hemophilia or Von Willebrand disease.
* No history of seizures within the last 3 months.
* No history of Lyme disease, unless six weeks' post treatment and no new symptoms, of Chagas disease, Babesiosis, or Leishmanias.
* Are not claustrophobic and are eligible to perform 3TMRI as per the MRI eligibility form.
* Do not have hip or knee replacements or other medical conditions that prevent 3TMRI research scans from being performed.

INCLUSION CRITERIA for the Non-Healthy-or-Frail and Frail groups:

* Age >= 20 years of age in the NHF group.
* Age >= 50 years of age in the F group.
* Are willing to return every 2 years for study visit procedures.
* Agree to genetic (DNA/RNA) sample collection, analysis, and storage.
* Have good venous access for blood sampling.
* Weigh >= 110lbs and a body mass index (BMI) <= 35.
* Do not have established genetic diseases such as sickle cell, hemochromatosis (iron overload), cystic fibrosis or Ehlers-Danlos syndrome (connective tissue disorder).
* Do not have important sensory deficits (legally blind and/or any condition that precludes the participant from being tested with standard neuropsychological tests or providing informed consent).
* Are able to read and speak English.
* Are able to understand the study risks and procedures, and consent to participate in the study.
* Not currently pregnant or a nursing mother.
* No current acute medical condition.
* No history of an active bleeding disorder such as hemophilia or Von Willebrand disease.
* No history of seizures within the last 3 months.
* Are not claustrophobic and are eligible to perform 3TMRI as per the MRI eligibility form.
* Do not have other medical conditions that prevent 3TMRI research scans from being performed.
* Frail participants meet the A and B criteria as reported.
* Not-Healthy-or-Frail participants will not be eligible for the Healthy group because of medical or functional problems and also do not meet the criteria for the Frail Group.

Participant Exclusion Criteria:

These criteria pertain to the Screening and Baseline Visits. If conditions considered as exclusion criteria for study entry develop any time after the Baseline evaluation, the participant remains in the study.

Exclusion Criteria:

* HIV virus infection (all groups).
* Hepatitis B or C (all groups).
* Active syphilis, gonorrhea or TB requiring treatment (all groups).
* WBC <3,000 or > 12,000/k/microL (only Healthy group).
* Platelets < 100,000 or >600,000 k/ microL (only Healthy group).
* Hemoglobin < 11.0 gm/dL in women and < 12.0 gm/dL in men (only Healthy group).
* GFR <50 mL/min/1.73 m^2 (only Healthy group)
* GFR <= to 30 (only non-Healthy-or-Frail group or Frail group)
* Bilirubin > 1.5 mg/dl (unless higher levels can be ascribed to Gilbert's disease (only Healthy group).
* ALT, AST, or alkaline phosphatase twice the normal serum concentration (only Healthy group).
* Corrected calcium < 8.5 or > 10.7 mg/dl (all groups).
* Albumin < 3.1 g/dl (only Healthy group).
* Cholesterol, LDL and/or Triglycerides >1.5x normal (only Healthy group).
* Positive Urine Drug Screen (unless taking prescribed medication and at the discretion of the PI) (all groups).
* Currently pregnant or a nursing mother (all groups).

Furthermore, if the participant is found eligible at Screening and Baseline but fails a urine drug screen (unless taking a prescribed medication and at the discretion of the PI) at any of the subsequent visits, the participant will be asked to return to repeat the test and if positive, will no longer be eligible to participate in the study.

Ages: 20 Years to 120 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy Volunteers, Non-Healthy/Non-Frail, Frail
Sampling Method: Probability Sample
Enrollment: 900 (Estimated)
Dates: Start 2015-03-15 (Actual); Primary Completion 2099-12-31 (Estimated); Study Completion 2099-12-31 (Estimated)

PRIMARY OUTCOMES:
Development of state-of-theart expression/methylation /protein PBMC atlas in aging | Ongoing
  measurement of epigenetic, gene expression, and protein biomarkers

CONTACTS AND LOCATIONS:
Overall Officials: Luigi Ferrucci, M.D., Principal Investigator — National Institute on Aging (NIA)
Locations (1):
- National Institute of Aging, Clinical Research Unit, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided
There is ongoing discussion within the NIA IRP and a plan has not been finalized yet.

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2015-AG-0063.html